CLINICAL TRIAL: NCT05364411
Title: HYpofractionated, Dose-redistributed RAdiotherapy With Protons and Photons to Combat Radiation-induced Immunosuppression in Head and Neck Squamous Cell Carcinoma (HYDRA)
Brief Title: HYpofractionated, Dose-redistributed RAdiotherapy With Protons and Photons in HNSCC
Acronym: HYDRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joris B.W. Elbers (Other)
Collaborators: Erasmus Medical Center (Other); HollandPTC (Industry)
Responsible Party: Sponsor-Investigator, Joris B.W. Elbers, Principal investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYDRA
Record Dates: First submitted 2022-04-28; First posted 2022-05-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Hypofractionation; Radiotherapy; Proton Therapy; Immune System Suppression
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Two parallel, non-comparative phase-I trials of HYDRA-protons run at HollandPTC (group 1, n=25) and HYDRA-photons (group 3, n=25) run at the Erasmus MC. Toxicity will be monitored until 1 year after the last patient has completed HYDRA. This will result in a median follow-up of approximately 2 years. Patients will subsequently receive follow-up according to standard of care up to 5 years after treatment for the evaluation of very late-onset toxicity.
  For translational immune profiling, HYDRA-protons and HYDRA-photons will be randomized by minimization (1:1 ratio) against SOC: conventional fractionated proton therapy in HPTC (group 2, n=25) and conventional fractionated photon therapy in the Erasmus MC (group 4, n=25), respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HYDRA-protons (Experimental): group 1, n=25, run at HollandPTC
  Interventions: Radiation: HYpofractionated, Dose-redistributed RAdiotherapy (HYDRA)
- Conventional fractionated proton therapy (Active Comparator): group 2, n=25, run at HollandPTC
  Interventions: Radiation: conventional fractionated radiotherapy
- HYDRA-photons (Experimental): group 3, n=25 run at Erasmus MC
  Interventions: Radiation: HYpofractionated, Dose-redistributed RAdiotherapy (HYDRA)
- Conventional fractionated photon therapy (Active Comparator): group 4, n=25 run at Erasmus MC
  Interventions: Radiation: conventional fractionated radiotherapy

INTERVENTIONS:
Radiation: HYpofractionated, Dose-redistributed RAdiotherapy (HYDRA) — 20 daily fractions, 5 times per week
  Arms: HYDRA-photons; HYDRA-protons
Radiation: conventional fractionated radiotherapy — 35 daily fractions, 5 times per week
  Arms: Conventional fractionated photon therapy; Conventional fractionated proton therapy

SUMMARY:
Radiotherapy for advanced-stage head and neck squamous cell carcinoma (HNSCC) results in an unfavorable 5-year overall survival of 40%, and there is a strong biological rationale for improving outcome by combinatorial treatment with immunotherapy. However, also immunosuppressive effects of radiotherapy have been reported and recently a randomized phase-III trial failed to show any survival benefit following the combination of a PD-L1 inhibitor with chemoradiotherapy. The hypothesis is that the combination of these individually effective treatments failed because of radiation-induced lymphodepletion and that the key therefore lies in reforming conventional radiotherapy, which typically consists of large lymphotoxic radiation fields of 35 fractions. By integrating modern radiobiology and individually established innovative radiotherapy concepts, the patient's immune system could be maximally retained. This will be achieved by 1) increasing the radiation dose per fraction so that the total number of fractions can be reduced (HYpofractionation), 2) by redistributing the radiation dose towards a higher peak dose within the tumor center and a lowered elective-field dose (Dose-redistribution) and 3) by using RAdiotherapy with protons instead of photons (HYDRA).

The objectives of this study are to determine the safety of HYDRA with protons and photons by conducting two parallel phase-I trials. HYDRA's efficacy will be compared to standard of care (SOC). The immune effects of HYDRA-protons will be evaluated by longitudinal immune profiling and compared to HYDRA-photons and SOC (with protons and photons). There will be a specific focus on actionable immune targets and their temporal patterns that can be tested in future hypofractionated-immunotherapy combination trials. This trial therefore is an important step towards future personalized immuno-radiotherapy combinations with the ultimate goal to improve survival for patients with HNSCC.

DETAILED DESCRIPTION:
The HYDRA dose prescriptions are, in 20 fractions (instead of the conventional 35 fractions):

* Inhomogeneous focal boost on the macroscopic gross tumor volume (GTVprimary tumor and GTVnodes) on FDG-PET: mean dose 59Gy, max dose 63Gy.
* The mean dose of 59Gy corresponds to an equal late normal tissue toxicity probability after conventionally fractionated radiotherapy of 70Gy in 35 fractions, considering an α/β=3 for normal tissue.
* Simultaneous integrated boost (SIB) on the clinical target volume (CTV-P1 = GTV+5mm): 55Gy
* Elective field / CTV-P2 (GTV+10mm): 40Gy

Patients who receive the HYDRA intervention treatment, as well as patients who receive standard of care may require the addition of a concurrent radiosensitizer based on clinicopathological features according to standard of care. Currently, the only two registered radiosensitizers are platinum-based chemotherapy (cisplatin/carboplatin) and cetuximab. These radiosensitizers should be administered according to standard care treatment protocols.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* ≥ 18 years old at time of signing informed consent.
* WHO 0-2
* Squamous cell carcinoma of the oropharynx, hypopharynx and larynx* proven by cytology / histology
* Patients amenable for curative intent proton therapy (by model-based selection criteria, according to the Dutch standard of care) or photon therapy.
* Radiotherapy with or without concurrent radiosensitizer.
* Ability to understand the requirements of the study and to give written informed consent, as determined by the treating physician.
* Written informed consent obtained.

  * Note: The HYDRA dose prescriptions should be applicable for all HNSCC patients and should therefore ideally be tested within the full range of treatment indications, e.g. multiple tumor subsites and both chemoradiotherapy and radiotherapy alone. There are several reports about acceptable acute toxicity following hypofractionated chemoradiotherapy in advanced stage HNSCC. However, concerns about late toxicity remain, especially for laryngeal carcinoma. Patients with laryngeal carcinoma are therefore initially excluded, until these patients are also considered eligible for treatment with HYDRA. The statistical considerations and interim safety analyses for this purpose and the decision-making / consultation are further described elsewhere.

Exclusion criteria

Patients who do not meet the inclusion criteria as specified in paragraph 4.2, and/or who meet the following additional criteria:

* Previously treated by irradiation on the same target volume
* Chronic inflammatory disease or immune disorders which, according to the principal investigator, may disturb the translational immune-read out.
* Patients currently under treatment for other malignant disease (unless in situ carcinoma or basal cell carcinoma of the skin), or treated for other malignant disease within the last 2 years.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule in the participating hospitals.
* Any other serious medical condition that could interfere with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety of HYDRA-protons and HYDRA-photons in terms of radiation-induced grade 3-4 late toxicity, physician-reported by CTCAE v5.0, monitored until 1 year after the last patient has completed HYDRA. | month 1-36
  HYDRA is randomized with standard of care for translational research purposes; a direct comparison of toxicity will statistically not be conclusive and is outside the scope of this study.

SECONDARY OUTCOMES:
Objective response after HYDRA defined by radiological response on CT-scans or MRI in comparison to standard of care | month 1-27
  Objective response rate 3 months after HYDRA (group 1 and 3), defined by radiological response on CT-scans or MRI using RECIST version 1.1 and/or histopathological confirmation of residual disease, in comparison to standard of care (group 2 and 4, respectively), 3 months after end of treatment
Efficacy of HYDRA in terms of in-field and nodal elective field tumor control at 1 year | month 24-36
  Efficacy of HYDRA (group 1 and 3) in terms of in-field and nodal elective field tumor control, 1 year after the last patient is included, in comparison to group 2 and 4, respectively.
Immune profile (changes) between all 4 treatment groups | month 1-27
  Numbers and phenotype of peripheral immune cell populations in blood at baseline, related to patient- and tumor characteristics, and differences between temporal changes of these immune markers during/after treatment at 6 timepoints in group 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Joris BW Elbers, MD, PhD, Principal Investigator — Erasmus MC, Rotterdam / HollandPTC, Delft - The Netherlands
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
tba

REFERENCES:
- [Derived] Elbers JBW, Gunsch PA, Debets R, Keereweer S, van Meerten E, Zindler J, van Norden Y, Hoogeman MS, Verduijn GM, Kroesen M, Nout RA. HYpofractionated, dose-redistributed RAdiotherapy with protons and photons to combat radiation-induced immunosuppression in head and neck squamous cell carcinoma: study protocol of the phase I HYDRA trial. BMC Cancer. 2023 Jun 13;23(1):541. doi: 10.1186/s12885-023-11031-w. PMID 37312053